CLINICAL TRIAL: NCT02513511
Title: Hypnosis as a Sole Agent to Perform Awake Intubation
Brief Title: Hypnosis to Perform Awake Intubation
Acronym: Hypnotube
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Patrick Schoettker,MD PD, MD, PD, University of Lausanne Hospitals
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 169/14
Record Dates: First submitted 2015-07-28; First posted 2015-07-31 (Estimated); Last update posted 2019-09-27 (Actual); Status verified 2019-09

CONDITIONS: Nasal Obstruction
Keywords: difficult airway; awake intubation
MeSH Terms: conditions — Nasal Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypnosis (Experimental): the investigators will put the patient into a hypnotic state and analyze laryngoscopy under hypnosis, followed by intubation.
  Interventions: Procedure: laryngoscopy under hypnosis

INTERVENTIONS:
Procedure: laryngoscopy under hypnosis — patient will be put in an hypnotic state before performing a laryngoscopy followed by oro-tracheal intubation

SUMMARY:
Awake intubation is a recommended safety procedure in specific cases where the intubation or ventilation before general anesthesia is at risk.

Numerous techniques to allow awake intubation have been described, such as pure awake technique, local anesthetics or intravenous sedation for example.

Hypnosis is used for various operating room techniques and surgeries. The investigators aim to analyze the feasibility of awake laryngoscopy and intubations on patients placed under hypnosis alone.

DETAILED DESCRIPTION:
Awake intubation is a recommended safety procedure in specific cases where the intubation or ventilation before general anesthesia is at risk.

Numerous techniques to allow awake intubation have been described, such as pure awake technique, local anesthetics or intravenous sedation for example.

Hypnosis is used for various operating room techniques and surgeries. The investigators aim to analyze the feasibility of awake laryngoscopy and intubations on patients placed under hypnosis alone.

Once patient will consent to be enrolled in the study, the same physician, trained in hypnosis, will accompany the patient in the operating room and place him into a hypnotic state. Once this hypnotic state is achieved, an oro-tracheal laryngoscopy will be performed with an Airtraq videolaryngoscope by an experienced anesthetist, specialised in the management of the difficult airway. If conditions allow it, the laryngoscopy will be followed by an oro-tracheal intubation.

A questionnaire assessing objective and subjective criteria from the patient and from the airway specialist will be collected.

ELIGIBILITY:
Inclusion Criteria:

* adults
* american society of anesthesiology classification 1-3
* understanding of french language

Exclusion Criteria:

* history of difficult intubation
* patient refusal
* deafness
* uncomfortable with french language understanding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2019-09-25 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Number of participants in which laryngoscopy is possible under hypnosis | 60 minutes
  laryngoscopy is feasible under hypnosis alone

SECONDARY OUTCOMES:
Number of participants in which intubation is possible under hypnosis | 60 minutes
  intubation is feasible under hypnosis alone
comfort assessed by patient | 60 minutes
  assessment of comfort on scale 1-5
comfort assessed by doctor | 60 minutes
  assessment of comfort on scale 1-5

CONTACTS AND LOCATIONS:
Overall Officials: patrick Schoettker, MD, PD, Principal Investigator — University of Lausanne Hospitals
Locations (1):
- Dpt of Anesthesiology, University of Lausanne CHUV, Lausanne, Canton of Vaud, Switzerland